CLINICAL TRIAL: NCT00942383
Title: Application of Novel, High Resolution, and Freehand Ultrasound Elasticity Imaging in Liver Surgery
Brief Title: Freehand Ultrasound Elasticity Imaging in Liver Surgery
Acronym: IOUS
Status: Terminated | Type: Observational
Why Stopped: low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Other Study IDs: J0765; NA_00011327 (Other: JHM IRB)
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2011-08

CONDITIONS: Liver Tumors
Keywords: liver tumor; liver tumors; liver cancer; hepatocellular carcinoma; metastatic colorectal cancer; metastatic cancer to the liver; metastatic cancer; metastatic neuroendocrine cancer; liver; liver surgery; radiofrequency ablation; microwave ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis; Carcinoma, Neuroendocrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IOUS-USEI: Receive intraoperative ultrasound (IOUS) using the Siemens Anteras to acquire ultrasound elasticity imaging (USEI) during standard of care surgical radiofrequency ablation and microwave ablation

SUMMARY:
The purpose of this study is to investigate the potential for visualizing radiofrequency-induced (RFA) and microwave-induced (MWA) hepatic thermal ablation lesions using a novel, high resolution, and freehand ultrasound elasticity imaging method in human subjects.

DETAILED DESCRIPTION:
Study Procedures This is a prospective cohort study. Data will be collected from patients who have signed an informed consent form and are undergoing open, laparoscopic, or percutaneous RFA or MWA as their treatment for liver tumors. Their images will be assembled and correlated according to their IOUS characteristics plus processed strain images. Below is the description of how each aim will be accomplished.

Aim-1: Ultrasound Elasticity Imaging Acquisition. USEI data (both raw US data and B-mode data) will be recorded during standard operative ultrasound imaging used to guide thermal ablative therapy in the operating room. Images will be acquired before, during, and after RFA or MWA therapy. Raw data acquisition will be conducted using a Siemens Antares US scanner (Siemens Medical Solutions USA, Inc. Ultrasound Division, Issaquah, WA) with an ultrasound research interface (URI) to access raw US data. A Siemens VF 10-5 linear array will be used to acquire data using manual handling. Typically, the ultrasound probe is tracked and spatially registered with the coordinate frame of the of the CT images, so the pixels of the B-mode images are known in the coordinate frame of the CT volume. Thus if one localizes the target anatomy in the B-mode images, then the position of the target is automatically known with respect to the CT volume for validation of the performance of the elastography. The tracking beams are standard B-mode pulses (6.67 MHz center frequency, F/1.5 focal configuration, apodized, pulse repetition frequency (PRF) of 10.6 KHz, with a pulse length of 0.3μs). This US device is one of the standard machines available for clinical US.

We will track the ultrasound probe with an Electro-Magnetic (EM) tracker. The tracker has small sensors that can be attached to the ultrasound probe under the sterile cover of the ultrasound probe, and therefore the sensor is not exposed. Also, the tracker has a 'transmitter' that is flat and is placed underneath the patient below a soft cushion. The sensor is attached to the ultrasound probe prior to the surgery and hencethe probe will remain sterile. The transmitter is flat and will be placed under a soft cushion so that it does not cause any pressure effects on patient.

In both cases (raw data and B-mode), the freehand acquisition should allow for palpation (manual compression within few millimeters). Risks and discomforts are negligible: Interventional ultrasound is FDA-approved, and we will use only the data resulting from standard of care use of clinically certified equipment. The maximum length of a data recording session will be 1-2 minutes during standard ultrasound acquisition. We will acquire cine sequences for five defined periods: 1) tumor imaging before probe placement; 2) immediately after probe placement; 3) near completion during ablation; 4) two minutes following ablation with probe in place; and 5) after removing the ablator probe.

ELIGIBILITY:
Inclusion Criteria:

* Any patient eligible for open, laparoscopic, or percutaneous hepatic RFA or MWA as their surgical treatment due to either primary tumors of the liver as well as liver metastases.
* Participants must be able to have post-operative CT/MRI at Johns Hopkins as their standard care.

Exclusion Criteria:

* Patients under 18 years old.
* Pregnant women.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing open, laparoscopic or percutaneous radiofrequency ablation (RFA) or microwave ablation (MWA) as treatment for liver tumors.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2012-06-13 (Actual); Study Completion 2012-06-13 (Actual)

PRIMARY OUTCOMES:
Comparison of transverse ablation diameter between intraoperative ultrasound elasticity imaging (USEI) and postoperative cross-sectional imaging (CT or MRI). | 2 years

SECONDARY OUTCOMES:
Comparison of ablation volume between ultrasound elasticity imaging (USEI) and CT/MRI. | 2 years
Correlation between "in vivo" versus phantom tumor size to validate the development of guidance systems combined with appropriate visualization and planning software for ablative therapy. | 2 years
Feasibility of image acquisition using Siemens Anteras clinical free-hand system. | 2 years
Feasibility of image processing and image segmentation using this clinical free-hand system. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Choti, M.D., Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- SKCCC, Baltimore, Maryland, United States